CLINICAL TRIAL: NCT07323576
Title: A Phase II, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of Inavolisib With Bevacizumab Plus Folfox or Folfiri as First Line Therapy in Patients With PIK3CA-Mutated Metastatic Colorectal Cancer
Brief Title: A Study to Evaluate the Efficacy and Safety of Inavolisib When Administered in Combination With Bevacizumab and FOLFOX or FOLFIRI as First Line Therapy in Participants With Colorectal Cancer
Acronym: INAVO-CRC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WO46300; 2025-523014-84-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-06; First posted 2026-01-07 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Cancer
Keywords: PIK3CA-mutated Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — inavolisib; Bevacizumab; Folfox protocol; IFL protocol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Randomized Period: FOLFOX or FOLFIRI + Bevacizumab + Inavolisib (Experimental): Participants will receive either FOLFOX or FOLFIRI and Bevacizumab along with Inavolisib.
  Interventions: Drug: Inavolisib; Drug: Bevacizumab; Drug: FOLFOX; Drug: FOLFIRI
- Randomized Period: FOLFOX or FOLFIRI + Bevacizumab + Placebo (Placebo Comparator): Participants will receive either FOLFOX or FOLFIRI and Bevacizumab along with Placebo.
  Interventions: Drug: Bevacizumab; Drug: FOLFOX; Drug: FOLFIRI; Drug: Placebo
- Safety Run-in Period: FOLFOX or FOLFIRI + Bevacizumab + Inavolisib (Experimental): Participants will receive either FOLFIRI or FOLFOX and Bevacizumab along with Inavolisib.
  Interventions: Drug: Inavolisib; Drug: Bevacizumab; Drug: FOLFOX; Drug: FOLFIRI

INTERVENTIONS:
Drug: Inavolisib — Participants will receive Inavolisib as per the schedule mentioned in the protocol.
  Other Names: Itovebi; GDC-0077
  Arms: Randomized Period: FOLFOX or FOLFIRI + Bevacizumab + Inavolisib; Safety Run-in Period: FOLFOX or FOLFIRI + Bevacizumab + Inavolisib
Drug: Bevacizumab — Participants will receive Bevacizumab as per the schedule mentioned in the protocol.
  Other Names: Avastin
Drug: FOLFOX — Participants will receive FOLFOX as per the schedule mentioned in the protocol.
Drug: FOLFIRI — Participants will receive FOLFIRI as per the schedule mentioned in the protocol.
Drug: Placebo — Participants will receive Placebo as per the schedule mentioned in the protocol.
  Arms: Randomized Period: FOLFOX or FOLFIRI + Bevacizumab + Placebo

SUMMARY:
This is a blinded Phase 2 study designed to evaluate the safety and efficacy of inavolisib with bevacizumab and chemotherapy, in participants with metastatic colorectal cancer (mCRC) whose tumors have a PIK3CA mutation. The study has a safety run-in period followed by a randomized period.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) <=1
* Histologically confirmed adenocarcinoma originating in the colon or rectum of the Stage 4 ( treatment plan does not include resection or curative ablation) per American Joint Committee on Cancer (AJCC) v8
* Measurable disease per RECIST v1.1
* No prior systemic therapy in the metastatic setting
* Confirmation of biomarker eligibility: documentation of a PIK3CA mutation from either central testing of tissue, or from a validated historically obtained (pre-existing) test of tumor tissue or blood may be used to confirm eligibility
* Adequate hematologic and organ function within 14 days prior to initiation of study treatment
* Agreement to adhere to the contraception requirements

Exclusion Criteria:

* Biomarker eligibility as per definition
* Type 2 diabetes requiring ongoing systemic treatment at the time of study entry or any history of Type 1 diabetes
* Residual Grade 2 or higher neuropathy due to prior oxaliplatin exposure (unless the participant is planned to be treated with FOLFIRI)
* Symptomatic, untreated, or actively progressing CNS metastases
* History of gastrointestinal (GI) fistula, GI perforation, or intra-abdominal abscess within 6 months prior to Day 1 of Cycle 1
* Treatment with strong cytochrome P450 (CYP) 3A4 inducers or strong CYP3A4 inhibitors within 1 week or 5 drug-elimination half-lives, whichever is longer, prior to initiation of study treatment (only for patients who will receive FOLFIRI)
* Known HIV positive status with exceptions for well controlled and on stable treatment
* History of malignancy within 5 years prior to screening, with the exception of the cancer under investigation in this study and malignancies with a negligible risk of metastasis or death

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
Safety Run-in Period: Percentage of Participants With Adverse Events (AEs) | Approximately 4 Years
Percentage of Participants With an Objective Response Rate | From Baseline Untill Radiographic Disease Progression (Approximately 4 Years)
  The percentage of participants with a confirmed complete response (CR) or confirmed partial response (PR) as determined by the investigator according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1.)

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | From Baseline Untill Radiographic Disease Progression (up to Approximately 4 Years)
  Time from randomization to death from any cause or the first occurrence of disease progression as determined by the investigator according to RECIST v1.1 (whichever occurs first)
Randomized Phase: Overall Survival (OS) | From Baseline Untill Death (up to Approximately 4 Years)
  Defined as the time from randomization to death from any cause
Randomized Phase: Disease Control Rate (DCR) | From Baseline Untill Disease Progression (up to Approximately 4 Years)
  Defined as the percentage of participants with stable disease for >=12 weeks or a CR or PR as determined by the investigator according to RECIST v1.1
Randomized Phase: Duration of Response (DOR) | From Baseline Untill Disease Progression or Death (up to Approximately 4 Years)
  Defined as the time from the first occurrence of a documented confirmed OR to death from any cause or the first occurrence of disease progression as determined by the investigator according to RECIST v1.1, (whichever occurs first)
Randomized Phase: Percentage of Participants With AEs | From Baseline up to 90 Days After the Final Dose of study treatment or Until Initiation of Another Anti-cancer Therapy (up to Approximately 4 Years)
Percentage of Participants With Symptomatic Treatment Toxicities as Assessed by National Cancer Institute Patient-Reported Outcomes Common Terminology Criteria for Adverse Events (NCI PRO-CTCAE) | Up to Approximately 4 Years
Percentage of Participants Troubled by Treatment Symptoms, as Assessed by Single Item European Organisation for Research and Treatment of Cancer Item Library 46 (EORTC IL46) | Up to Approximately 4 Years
Change From Baseline in Symptomatic Treatment Toxicities as Assessed by PRO-CTCAE | Baseline up to Approximately 4 Years
Change From Baseline in Treatment Side-effect Bother as Assessed by EORTC IL46 item | Baseline up to Approximately 4 Years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing